CLINICAL TRIAL: NCT07078331
Title: A Prospective, Multi Center, Single-Blinded, Randomized, Controlled Study to Evaluate the Safety and Performance, and Dose, of OsteoAdapt DE in Localized Alveolar Ridge Augmentations for Defects Associated With Extraction Sockets - Feasibility Study
Brief Title: Safety and Performance, and Dose, of OsteoAdapt DE in Localized Alveolar Ridge Augmentations
Acronym: RESTORE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theradaptive, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: OADE.D1.ISR
Record Dates: First submitted 2025-07-09; First posted 2025-07-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Tooth Extraction Site Healing; Ridge Augmentation; Bone Graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The Subjects will be blinded to their arm allocation whereas the treating physician will be unblinded (Single blinded study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Low Dose OsteoAdapt DE (Experimental): OsteoAdapt DE with 0.8 mg AMP2 per cc of ReBOSSIS-J packed inside of the extraction socket
  Interventions: Device: OsteoAdapt DE (0.8 mg)
- High Dose OsteoAdapt DE (Experimental): OsteoAdapt DE with 2.0 mg AMP2 per cc of ReBOSSIS-J packed inside of the extraction socket
  Interventions: Device: OsteoAdapt DE (2.0 mg)
- Control (Xenograft) (Active Comparator): Xenograft particulate bone graft packed inside of the extraction socket (SOC).
  Interventions: Device: Xenograft Bone Graft

INTERVENTIONS:
Device: OsteoAdapt DE (0.8 mg) — Procedure of single tooth extraction and grafting along with related data collection:
  Implanted OsteoAdapt DE bone graft (0.8 mg) by a trained and qualified study investigator per the IFU, IB and CIP guidelines
  Arms: Low Dose OsteoAdapt DE
Device: OsteoAdapt DE (2.0 mg) — Procedure of single tooth extraction and grafting along with related data collection:
  Implanted OsteoAdapt DE bone graft (2.0 mg) by a trained and qualified study investigator per the IFU, IB and CIP guidelines
  Arms: High Dose OsteoAdapt DE
Device: Xenograft Bone Graft — Procedure of single tooth extraction and grafting along with related data collection:
  Implanted xenograft bone graft by a trained and qualified study investigator per the IFU, IB and CIP guidelines
  Arms: Control (Xenograft)

SUMMARY:
This study's objective is to evaluate OsteoAdapt DE's safety and performance in comparison to Xenograft particulate bone graft for alveolar ridge augmentation. Additionally, the study aims to optimize OsteoAdapt DE dosing for future studies by assessing two concentrations: a low dose (0.8 mg/cc) and a high dose (2.0 mg/cc).

DETAILED DESCRIPTION:
Prospective, Multi Center, Single-Blinded, Randomized, Controlled Study to Evaluate the Safety and Performance, and Dose, of OsteoAdapt DE in Localized Alveolar Ridge Augmentations for Defects Associated with Extraction Sockets - Feasibility Study.

Patients requiring a single tooth extraction (with the intent of placing a dental implant into the regenerated bone in the extraction socket) who signed the consent form and are found eligible for the study (meet the inclusion criteria and none of the exclusion criteria) will be randomized into one of 3 study Arms at a 1:1:1 ratio prior to the extraction procedure:

Study Arm 1 - Investigational (~15 subjects): OsteoAdapt DE with 0.8mg AMP-2 per cc of ReBOSSIS-J packed inside of the extraction socket.

Study Arm 2 - Investigational (~15 subjects): OsteoAdapt DE with 2.0mg AMP2 per cc of ReBOSSIS-J packed inside of the extraction socket.

Study Arm 3 - Control (~15 subjects): Xenograft particulate bone graft packed inside of the extraction socket (SOC).

The Subjects will be blinded to their arm allocation whereas the treating physician will be unblinded (Single blinded study). Grafting of the prepared socket will be performed at the time of tooth extraction, and all extraction sockets will be covered with a resorbable collagen membrane (e.g. BioGide from Geistlich) prior to reapproximation of buccal and lingual flaps. Primary closure of the extraction socket is not required.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 or older at the time of signing informed consent
2. Subject requires extraction of a single tooth due to extensive carious lesions, prosthetic or endodontic failure, root fracture, or other reasons with dental implant treatment planned at the site
3. Tooth root in position allowing a bone core sample to be harvested within the former socket
4. 6mm of alveolar bone height without impinging on the maxillary sinus or inferior alveolar canal
5. Dehiscence of ≤ 2 mm on the buccal bony wall at the time of extraction
6. Presence of other socket walls, mesial, distal and lingual walls
7. The subject is willing and able to be present for routine follow up visits, comply with postoperative management program, and is able to understand and sign the informed consent form
8. Willing to use a reliable method of contraception (for woman of childbearing potential and males with a partner who is of childbearing potential)

Exclusion Criteria:

1. Active localized or systemic infection
2. Untreated periodontal disease
3. Presence of a fenestration larger than 3 mm in diameter in the buccal wall at the time of extraction
4. Inadequate bone dimensions or restorative space to place a dental implant
5. The subject uses, or has used within 30 45 days of surgery, tobacco or nicotine or is prescribed steroids such as cortisone
6. Presence or history of malignancy (excludes surgically resected skin squamous cell or basal cell carcinoma), radiotherapy, or chemotherapy for any malignancy within the last 5 years. History of malignancy may include multiple exostoses syndrome (also known as multiple osteochondromas syndrome), an inherited condition associated with bumps of cartilage on the bones, which has been associated with an increased risk of chondrosarcoma); individuals with hereditary cancer syndromes are excluded. Examples of hereditary cancer syndromes are hereditary breast and ovarian cancer syndrome, Li-Fraumeni syndrome, Cowden syndrome, and Lynch syndrome. Also called family cancer syndrome and inherited cancer syndrome individuals who have undergone any transplant surgery and are on immunosuppressant therapy
7. Has a history of any endocrine or metabolic disorder known to affect osteogenesis (e.g.: Paget's disease, renal osteodystrophy, Ehler-Danlos syndrome, or osteogenesis imperfecta)
8. Insulin dependent diabetes
9. History of exposure to any recombinant proteins or peptides used for bone formation (i.e., Infuse Bone Graft, AUGMENT Bone Graft, GEM21S, i-FACTOR Peptide Enhanced Bone Graft, or PepGen P-15 Synthetic Bone Graft)
10. Hypersensitivity or allergy to any components of the study treatments including, but not limited to, bone morphogenetic proteins (BMPs); tricalcium phosphate (TCP); PLGA polymer
11. History of any allergy resulting in anaphylaxis
12. Treatment with an investigational therapy (drug, device, and/or biologic) within 120 days (or 5 half-lives, whichever is greater) prior to implantation surgery, or such treatment is planned during the 24-month period following implantation of the study treatment; prior or planned use of rhBMP-2
13. Pregnant at final Screening evaluation prior to Day 1 pre-procedure or interested in trying to conceive a child (both females and males) in the next 12 months or nursing
14. Any condition that would interfere with the subject's ability to comply with study instructions or prohibit Radiographic assessments that might confound the interpretation of the study or put the subject at risk
15. Patients taking any drug known to interfere with bone/soft tissue healing. See "Medication protocol" section of the protocol.
16. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful placement of a dental implant with primary stability (>25 N cm) | 6 months
Rates of serious adverse events related to the grafting material and / or grafting procedure | 6 months
Occurrence of any unplanned additional procedures at the implantation site related to the grafting material or grafting procedure | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- Armenia (2):
  - Armenia Medical Center, Yerevan
  - Medline Clinic, Yerevan
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Assuta Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky